CLINICAL TRIAL: NCT04312438
Title: Safety of Oral Food Challenge With Cow's Milk Proteins in Children With Food Allergy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Tatiana Jamer, Principal Inverstigator, Wroclaw Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OFC2020
Record Dates: First submitted 2020-03-08; First posted 2020-03-18 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Food Allergy
Keywords: oral food challenge; food allergy; children
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 13 mo to 15 yo children diagnosed with Cow's Milk Allergy (Experimental): oral food challenge with cow's milk proteins
  Interventions: Diagnostic Test: oral food challenge with cow's milk proteins

INTERVENTIONS:
Diagnostic Test: oral food challenge with cow's milk proteins — in children with diagnosed Cow's Milk Allergy open oral food challenge test with cow's milk protein (milk formula in children up to 3 yo, cow,s milk after 3 yo) will be carried out

SUMMARY:
The aim of the study is to assess the safety of an oral food challenge (OFC) with cow's milk proteins and to assess the tolerance of cow's milk proteins in children with a food allergy after introducing cow's milk into the diet.

DETAILED DESCRIPTION:
The aim of the study is to assess the safety of an oral food challenge test with cow's milk proteins and to assess the tolerance of cow's milk proteins in children with food allergies after introducing cow's milk into the diet.

The study covers children over 12 months of age diagnosed with cow's milk allergy, treated with a non-dairy elimination diet based on extensively-hydrolyzed formulas or amino acid formulas, admitted to the Department of Pediatrics, Gastroenterology and Nutrition to conduct an open oral food challenge. In all children, after appropriate assessment and qualification (interview, physical examination, skin prick tests, results of allergen - specific immunoglobulin E (IgE), total blood count, fecal calprotectin and lactoferrin), an oral food challenge test with cow's milk will be performed. The oral food challenge test will be carried out in accordance with current standards and with child protection in the event of an adverse reactions. During the food challenge test (first 24 hours), after 2 weeks (phone survey) and 3 months after the test (visit to the Department) the frequency, severity and type of allergic reactions and cow's milk protein tolerance will be assessed. The safety of oral food challenge with cow's milk protein in children previously fed with extensively - hydrolyzed formulas or amino acid formulas will be compared. The results of allergy tests, total blood count and intestinal inflammatory markers (fecal calprotectin and fecal lactoferrin) will also be assessed before and 12 weeks after oral food challenge. The assessment of the incidence and severity of allergic reactions and tolerance of cow's milk proteins after introduction into the diet in children challenged with cow's milk proteins may help to establish guidelines on the qualifications and how to conduct an oral challenge test.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 13 months to 15 years
* children diagnosed with cow's milk allergy treated with a dairy-free diet
* informed consent of the child's parents/legal guardians to participate in the study

Exclusion Criteria:

* occurrence of anaphylactic reaction after ingestion cow's milk proteins less than 12 months
* positive skin prick test with cow's milk proteins
* milk specific serum IgE values > 17,5 kU/L
* age below 13 moths
* no consent of the child's parents/legal guardians to participate in the study

Ages: 13 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of allergic reaction during and after oral food challenge assessed by the occurrence of allergic symptoms in children | up to 12 weeks after oral food challenge
  assessment of type, severity and frequency of food allergy symptoms (allergic skin changes, gastrointestinal and respiratory tract symptoms) that occurred during and after oral food challenge, based on medical history data and physical examination collected by a doctor
Change of hemoglobin level after 12 weeks after oral food challenge | before and 12 weeks after oral food challenge
  hemoglobin concentration in venous blood measured in g/dl
Changes in skin prick test results 12 weeks after oral food challenge | before and 12 weeks after oral food challenge
  skin prick test with milk, egg yolk, egg white, chicken, wheat, fish before and 12 weeks after oral food challenge
Changes in allergen - specific IgE pediatric panel results 12 weeks after oral food challenge | before and 12 weeks after oral food challenge
  allergen - specific IgE pediatric panel results (allergen - specific IgE concentration measured in kU/l, classified in grades 0-6) before and 12 weeks after oral food challenge
Change of fecal calprotectin concentrations (intestinal inflammatory marker) after 12 weeks after oral food challenge | before and 12 weeks after oral food challenge
  concentration of fecal calprotectin in the feces measured in ug/g before and 12 weeks afte oral food challenge
Change of fecal lactoferrin concentrations (intestinal inflammatory marker) after 12 weeks after oral food challenge | before and 12 weeks after oral food challenge
  concentration of fecal lactoferrin in the feces measured in μg/g before and 12 weeks afte oral food challenge

SECONDARY OUTCOMES:
Comparison of the incidence of allergic reaction during and after oral food challenge with cow's milk protein between children previously fed with extensively - hydrolyzed formulas and amino acid formulas | up to 12 weeks after oral food challenge
  assessment of type, severity and frequency of food allergy symptoms (allergic skin changes, gastrointestinal and respiratory tract symptoms) that occurred during and after oral food challenge, based on medical history data and physical examination collected by a doctor
Comparison of changes in skin prick test results between children previously fed with extensively - hydrolyzed formulas and amino acid formulas | before and 12 weeks after oral food challenge
  skin prick test with milk, egg yolk, egg white, chicken, wheat, fish before and 12 weeks after oral food challenge
comparison of changes in allergen - specific IgE pediatric panel results between children previously fed with extensively - hydrolyzed formulas and amino acid formulas | before and 12 weeks after oral food challenge
  allergen - specific IgE pediatric panel results (allergen - specific IgE concentration measured in kU/l, classified in grades 0-6) before and 12 weeks after oral food

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Jamer, PhD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

REFERENCES:
- [Background] Muraro A, Werfel T, Hoffmann-Sommergruber K, Roberts G, Beyer K, Bindslev-Jensen C, Cardona V, Dubois A, duToit G, Eigenmann P, Fernandez Rivas M, Halken S, Hickstein L, Host A, Knol E, Lack G, Marchisotto MJ, Niggemann B, Nwaru BI, Papadopoulos NG, Poulsen LK, Santos AF, Skypala I, Schoepfer A, Van Ree R, Venter C, Worm M, Vlieg-Boerstra B, Panesar S, de Silva D, Soares-Weiser K, Sheikh A, Ballmer-Weber BK, Nilsson C, de Jong NW, Akdis CA; EAACI Food Allergy and Anaphylaxis Guidelines Group. EAACI food allergy and anaphylaxis guidelines: diagnosis and management of food allergy. Allergy. 2014 Aug;69(8):1008-25. doi: 10.1111/all.12429. Epub 2014 Jun 9. PMID 24909706
- [Background] Roberts G. Food challenges, the risks and benefits. Clin Exp Allergy. 2017 Sep;47(9):1106-1107. doi: 10.1111/cea.12999. No abstract available. PMID 28856837
- [Background] Beigelman A. To Eat or Not to Eat? Introduction of Food After Negative Oral Food Challenge. J Allergy Clin Immunol Pract. 2017 Mar-Apr;5(2):477-478. doi: 10.1016/j.jaip.2016.09.005. No abstract available. PMID 28283161
- [Background] Nowak-Wegrzyn A, Assa'ad AH, Bahna SL, Bock SA, Sicherer SH, Teuber SS; Adverse Reactions to Food Committee of American Academy of Allergy, Asthma & Immunology. Work Group report: oral food challenge testing. J Allergy Clin Immunol. 2009 Jun;123(6 Suppl):S365-83. doi: 10.1016/j.jaci.2009.03.042. PMID 19500710
- [Background] Cox AL, Nowak-Wegrzyn A. Innovation in Food Challenge Tests for Food Allergy. Curr Allergy Asthma Rep. 2018 Oct 30;18(12):74. doi: 10.1007/s11882-018-0825-3. PMID 30377836
- [Background] Gupta M, Cox A, Nowak-Wegrzyn A, Wang J. Diagnosis of Food Allergy. Immunol Allergy Clin North Am. 2018 Feb;38(1):39-52. doi: 10.1016/j.iac.2017.09.004. Epub 2017 Oct 23. PMID 29132673